CLINICAL TRIAL: NCT01134601
Title: A Phase I Study of AZD6244 in Combination With Capecitabine and Radiotherapy in Locally Advanced Adenocarcinoma of the Rectum
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: As per Cancer Therapy Evaluation Program (CTEP), this protocol has only enrolled one participant and it is unlikely that the study will be able to be completed successfully. CTEP slated the protocol to be administratively closed.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100132; 10-C-0132
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Non-Metastatic Adenocarcinoma of the Rectum
Keywords: Rectal Cancer; Radiation Therapy; Capecitabine; AZD6244
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Capecitabine; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2 (Experimental): LEVEL 1 - Cycle = 49 days: AZD6244: 50 mg by mouth (PO) everyday (QD) Capecitabine: 825 mg/m^2 by mouth (PO)
  Interventions: Procedure: Radiation Therapy; Drug: Capecitabine; Drug: AZD6244

INTERVENTIONS:
Procedure: Radiation Therapy
Drug: Capecitabine
  Other Names: Xeloda
Drug: AZD6244
  Other Names: Selumetinib

SUMMARY:
Background:

- The investigational anti-cancer drug Selumetinib (AZD6244) prevents a protein found in rectal cancer from working properly, which may slow tumor growth and allow radiation and chemotherapy treatments to destroy more cancer cells. Researchers are interested in determining whether AZD6244 can be used to improve treatment outcomes in individuals who have rectal cancer that has spread outside the rectum into the surrounding pelvis.

Objectives:

- To determine safe and effective doses of AZD6244, along with radiation and chemotherapy, to treat rectal cancer.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with rectal cancer that has spread outside the inner wall of the rectum or into lymph nodes in the pelvis.

Design:

* Eligible participants will be screened with a physical examination, blood and tumor samples, and imaging studies.
* Participants will receive AZD6244 twice a day by mouth for 1 full week (7 days) before starting radiation and chemotherapy and every week thereafter until the end of the radiation and chemotherapy treatment.
* Participants will have radiation therapy daily, 5 days per week, for approximately 6 weeks.
* Participants will receive chemotherapy (capecitabine) twice daily, 5 days per week, for approximately 6 weeks.
* Approximately 4 to 8 weeks after completing the AZD6244, radiation, and chemotherapy treatment, participants may have surgery to remove any tumors and affected lymph nodes. This surgery is not part of the treatment delivered on this protocol.
* Participants will have a follow-up exam 3 weeks after the end of treatment, every 3 months for the first year, and then in the second and third year after the end of treatment. These visits will involve a full medical examination and imaging studies.

DETAILED DESCRIPTION:
Background:

* Local recurrences of rectal cancer are morbid and difficult to manage effectively.
* Colorectal cancers frequently harbor rat sarcoma (RAS) mutations and Epidermal growth factor (EGF)/epidermal growth factor receptor (EGFR) over-expression.
* AZD6244 is an orally available selective, adenosine triphosphate uncompetitive inhibitor of methyl ethyl ketone (MEK)1/2 that sensitizes tumor cells to radiation in vitro and in vivo.

Objectives:

Primary

* To define the maximum tolerable dose of AZD6244 Hyd-Sulfate delivered twice a day (BID), 7 days per week, in combination with radiation therapy (RT) and Capecitabine in patients with locally advanced adenocarcinoma of the rectum without distant metastases.
* To define the dose-limiting toxicities and toxicity profile associated with administration of AZD6244 Hyd-Sulfate delivered BID, 7 days per week in combination with RT and Capecitabine

Secondary

* To evaluate the pharmacokinetics of AZD6244 delivered alone and in combination with Capecitabine 825 mg/m(2) by mouth (PO) BID.
* To obtain exploratory information regarding the pathologic response rate obtained after treatment with the maximum tolerated dose (MTD) of AZD6244 Hyd-Sulfate in combination with Capecitabine and 50.4 Gray (Gy) of RT.
* To determine if changes in phosphorylated extracellular-signal regulated kinase (ERK) (pERK) in peripheral blood mononuclear cells correlates to changes in phosphorylated extracellular-signal regulated kinase (pERK) in rectal tumors in the setting of treatment with AZD6244.
* To perform an exploratory analysis to determine if the presence of activating mutations in RAS or BRAF in tumor or changes in plasma transforming growth factor-alpha (TGFalpha) levels and tumor pERK/total ERK with AZD6244 treatment alone and after AZD6244 in combination with Capecitabine and RT predicts for down staging or pathologic response.

Eligibility:

* Histologically or cytologically confirmed locally advanced, non-metastatic adenocarcinoma of the rectum (clinical stage T3AnyN, T4AnyN, or AnyTN+).
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Normal organ and marrow function.

Design:

* All patients will receive 50.4 Gy of RT to the pelvis and rectal tumor delivered concurrently with Capecitabine and AZD6244. AZD6244 will be delivered BID daily, 7 days per week, in a dose escalated fashion. AZD6244 will begin one week prior to Capecitabine and RT and will conclude on the last day of Capecitabine and RT.
* Capecitabine will be delivered at 825 mg/m(2) PO every 12 hours, 5 days per week, starting on the first day of RT and continuing until the last day of RT.
* Biopsies of tumor tissue will be obtained prior to treatment, after one week of AZD6244, and after one week of AZD6244, RT, and Capecitabine for correlative assays.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed locally advanced, non-metastatic adenocarcinoma of the rectum (clinical stage T3 anyN, T4 anyN, or AnyT N+).
* Patients with recurrent adenocarcinoma of the rectum with no clinically evident distant disease will be eligible if they are deemed to have pelvic nodal metastases or disease extending through the muscularis of the rectum. These patients should be evaluated by a Radiation Oncologist, Medical Oncologist and Surgeon prior to enrolling on study to confirm anticipated resectability. These patients should not have received prior radiotherapy for management of their rectal cancer.
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 70%).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets: greater than or equal to 100,000/mcL
  * total bilirubin: within normal institutional limits except for patients with Gilbert's who must have a direct bilirubin of less than 1.0 mg/dL
  * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times the institutional upper limit of normal
  * creatinine within normal institutional limits

OR

-- creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for six months after the completion of radiation. Women of child-bearing potential must have a negative pregnancy test prior to entry. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Adequate contraception for male patients should be used for 6 months after irradiation.
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to sign a release of medical records pertaining to previous and future treatment for rectal cancer.

EXCLUSION CRITERIA:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or lack of recovery from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 or other agents used in study.
* Previous methyl ethyl ketone (MEK) inhibitor use.
* Contraindications to radiotherapy to the pelvis such as inflammatory bowel disease or known genetic sensitivity to ionizing radiation such as ataxia telangiectasia.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with corrected QT interval (QTc) interval greater than 470 msecs or other factors that increase the risk of Q wave, T wave (QT) prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class III and IV definitions are excluded.
* Required use of a concomitant medication that can prolong the QT interval. A comprehensive list of agents with the potential to cause QTc prolongation can be found at http://www.arizonacert.org/medical-pros/drug-lists/drug-lists.htm.
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy.
* Known dihydropyrimidine dehydrogenase deficiency.
* History of prior radiation to the pelvis
* For patients with newly diagnosed rectal cancer, prior therapy for adenocarcinoma of the rectum with the exception of diverting colostomy if required to relieve obstruction (including chemotherapy).
* Patients with recurrent rectal cancer may not have undergone prior radiotherapy for rectal adenocarcinoma or have received therapy for the recurrence with the exception of diverting colostomy if required to relieve obstruction.
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* Uncontrolled hypertension
* Pregnant or lactating females are excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05-24 (Actual); Primary Completion 2012-10-22 (Actual); Study Completion 2012-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies BR, Logie A, McKay JS, Martin P, Steele S, Jenkins R, Cockerill M, Cartlidge S, Smith PD. AZD6244 (ARRY-142886), a potent inhibitor of mitogen-activated protein kinase/extracellular signal-regulated kinase kinase 1/2 kinases: mechanism of action in vivo, pharmacokinetic/pharmacodynamic relationship, and potential for combination in preclinical models. Mol Cancer Ther. 2007 Aug;6(8):2209-19. doi: 10.1158/1535-7163.MCT-07-0231. PMID 17699718
- [Background] O'Neill E, Kolch W. Conferring specificity on the ubiquitous Raf/MEK signalling pathway. Br J Cancer. 2004 Jan 26;90(2):283-8. doi: 10.1038/sj.bjc.6601488. PMID 14735164
- [Background] Wellbrock C, Ogilvie L, Hedley D, Karasarides M, Martin J, Niculescu-Duvaz D, Springer CJ, Marais R. V599EB-RAF is an oncogene in melanocytes. Cancer Res. 2004 Apr 1;64(7):2338-42. doi: 10.1158/0008-5472.can-03-3433. PMID 15059882

RESULTS

PARTICIPANT FLOW:
Groups:
- Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2: LEVEL 1 - Cycle = 49 days: AZD6244: 50 mg by mouth (PO) everyday (QD) Capecitabine: 825 mg/m^2 by mouth (PO)
  Radiation Therapy
  Capecitabine
  AZD6244
Period: Overall Study
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerable Dose of Selumetinib (AZD6244) Hyd-Sulfate in Combination With Radiation Therapy (RT) and Capecitabine in Participants With Locally Advanced Adenocarcinoma of the Rectum.
Description: Maximum tolerable dose is defined as the dose level at which no more than 1 of 6 participants experience dose limiting toxicity (DLT) during treatment and the three weeks after completion. Examples of DLT is recurring and persistent Grade 3 diarrhea despite appropriate medical therapy, absolute neutrophil count <500 for more than 5 days or neutropenic fever, Grade 3 thrombocytopenia, Grade 4 fatigue, and Grade 4 dermatitis acneiform rash.
Time Frame: During treatment and within first 3 weeks after treatment
Population: This outcome measure was not done. As per the Cancer Therapy Evaluation Program (CTEP), this protocol has only enrolled one participant and it is unlikely that the study will be able to be completed successfully. CTEP slated the protocol to be administratively closed.
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 0

2. Secondary Outcome: Pharmacokinetics of Selumetinib (AZD6244) in Combination With Capecitabine
Description: To evaluate the pharmacokinetics of AZD6244 in Combination with Capecitabine using logistic regression.
Time Frame: Pre-and post treatment
Population: as for outcome 1
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Phosphorylated ERK (pERK) in Peripheral Blood Mononuclear Cells and Tumor, and Transforming Growth Factor Alpha (TGFa) Levels
Description: Changes in phosphorylated ERK (pERK) in peripheral blood mononuclear cells and tumor, and TGFa levels measured by flow cytometry.
Time Frame: Pre-and post treatment
Population: as for outcome 1
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Here is the Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, and up to 30 days following the last dose of study drug, approximately 14 months and 26 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 1
Participants | 1

5. Other Pre Specified Outcome: Pathologic Complete Response Rate
Description: To obtain exploratory information regarding the pathologic response rate. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Complete Response is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: After treatment with the maximum tolerated dose
Population: as for outcome 1
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Dose-Limiting Toxicity (DLT)
Description: Examples of DLT is recurring and persistent Grade 3 diarrhea despite appropriate medical therapy, absolute neutrophil count <500 for more than 5 days or neutropenic fever, Grade 3 thrombocytopenia, Grade 4 fatigue, and Grade 4 dermatitis acneiform rash.
Time Frame: During treatment and within first 3 weeks after treatment
Population: as for outcome 1
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, and up to 30 days following the last dose of study drug, approximately 14 months and 26 days.
Arm/Group | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib (AZD6244): 50 mg & Capecitabine: 825 mg/m^2 (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (3)
CPK increased (Investigations) | 1 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (3)
Lymphocyte count increased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, perianal erythema (Skin and subcutaneous tissue disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-10-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT01134601/Prot_SAP_000.pdf
  • Informed Consent Form (2011-10-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT01134601/ICF_001.pdf